CLINICAL TRIAL: NCT02435420
Title: A Retro-prospective Study of Total Hip Arthroplasty With EMPERION Modular Primary Stem in Australian Centres
Brief Title: A Retro-prospective Study of Total Hip Arthroplasty With EMPERION Modular Primary Stem in Australian Centres (HISTORIC)
Acronym: HISTORIC
Status: Terminated | Type: Observational
Why Stopped: Commercial decision
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-4542-03
Record Dates: First submitted 2015-04-30; First posted 2015-05-06 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Osteoarthritis, Hip; Arthritis, Degenerative
Keywords: Total Hip Arthroplasty; EMPERION Modular Stem; Survivorship
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EMPERION Modular Primary Stem subjects: All subjects have previously been implanted with the EMPERION Modular Primary Stem for primary total hip arthroplasty.
  Interventions: Device: EMPERION Modular Primary Stem

INTERVENTIONS:
Device: EMPERION Modular Primary Stem — Primary total hip arthroplasty using the EMPERION Modular Primary Stem

SUMMARY:
This is a retro-prospective, single arm, sequential enrolment study to collect relevant clinical and radiological data in at least 156 subjects, at up to 10 sites in Australia, who have been implanted with the EMPERION™ Modular Hip System in primary THA procedures to assess its safety and efficacy over 5 years post-surgery.

DETAILED DESCRIPTION:
The main aim of the study is to demonstrate that there is no significant difference in survivorship at 5 years in the EMPERION™ primary stem compared to other primary stems for total hip arthroplasty.

Investigational site personnel will review and screen clinical records for potential subjects to be included in the study. Eligible patients will be contacted and follow-up status and implant revision status will be assessed at this initial contact. The subject will be given the option to participate in a prospective 5-year on-site follow-up visit for which they will provide written informed consent. An HREC waiver of informed consent for study participation will be obtained for subjects who are lost to follow-up, deceased or are unwilling/unable to participate in a prospective on-site 5-year follow-up visit, allowing the inclusion of data from all patients implanted with the study device regardless of follow-up status and therefore eliminate selection bias.

Data will be collected retrospectively from the subject pre-surgery, during surgery, at discharge and at 1-year follow-up found in their medical files and prospective data will be collected from the subject's 5-year Follow-up visit and documented on specially designed Case Report Forms (CRFs).

Data to be collected include:

* Subject demographics
* Primary diagnosis for THA
* Additional relevant history and physical findings
* Post-operative follow-up findings at 1 and 5 years
* Radiological Assessment
* Revision by time points
* Adverse Events

ELIGIBILITY:
Inclusion Criteria:

1) Subject has undergone primary total hip arthroplasty with the EMPERION™ Modular hip system

Exclusion Criteria:

1. Subject received the EMPERION™ THA on the affected hip as a revision for a previously failed THA
2. At the time of surgery, subject had an active infection or sepsis (treated or untreated)
3. At the time of surgery, subject had presence of malignant tumor, metastatic or neoplastic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects that have been implanted with the EMPERION modular primary stem for primary total hip arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Survivorship of stem | 5 years

SECONDARY OUTCOMES:
Revision for any reason | 5 years
Radiographic Assessment | 5 years
  Radiographic problems, component orientation, radiolucencies, migration, osteolysis, stress shielding, subsidence
Harris Hip Score | 5 years
Adverse Events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr David Liu, BSc, M.B., B.S. F, Principal Investigator — John Flynn Private Hospital
Locations (8):
- Australia (8):
  - Dubbo Base Hospital, Dubbo, New South Wales
  - Dubbo Private Hospital, Dubbo, New South Wales
  - North Shore Private Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Hip and Knee Clinic at Sydney Olympic Park, Sydney, New South Wales
  - Mater Health Services, South Brisbane, Queensland
  - John Flynn Hospital, Tugun, Queensland
  - Epworth Centre, Melbourne, Victoria